CLINICAL TRIAL: NCT01402557
Title: Telehealth for Weight Maintenance of African-American Women
Brief Title: Telehealth for Weight Maintenance of African-American Women ("Exercise Your Faith")
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ben Gerber, Professor of Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2006-0836; R21DK078352 (NIH)
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Overweight; Obesity
Keywords: Obesity; Body Weight Changes; Internet
MeSH Terms: conditions — Overweight; Obesity; Body Weight Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telephone Support Only (Active Comparator): These participants receive telephone support only during the weight maintenance phase.
  Interventions: Behavioral: Weight Loss Church Program; Behavioral: Telephone Counseling
- Telehealth (Experimental): These participants receive telehealth support (with Internet-enabled digital video recorders) during the weight maintenance phase. These participants also receive telephone support monthly.
  Interventions: Behavioral: Weight Loss Church Program; Behavioral: Telephone Counseling; Behavioral: Telehealth Support

INTERVENTIONS:
Behavioral: Weight Loss Church Program — An initial 12-week weight loss program held in churches to ensure adequate participation, competence in performing exercises, and development of social relationships among participants. All participants attend the church programs prior to the weight maintenance phase.
Behavioral: Telephone Counseling — Following completion of the weight loss program, participants will receive monthly telephone counseling.
Behavioral: Telehealth Support — After the weight loss program, women will access the home weight maintenance telehealth program through Internet enabled digital video recorders connected to their television sets. The telehealth program includes three components: (1) Weekly Video: home access to weekly video programs including problem solving and relapse prevention strategies, as well as motivational stories; (2) Teleexercise: home access to updated video exercise programs; and (3) Electronic Communication: social support through online communication with other participants, and with an exercise and nutrition interventionist.
  Arms: Telehealth

SUMMARY:
Obesity can cause many health problems, including high blood pressure, diabetes, heart disease, and stroke. Although some people may lose weight through diet and exercise, many regain weight over time. There is a need to study new ways of helping people maintain their weight. The purpose of this research is to study the effect of a weight maintenance program provided through home television sets connected to the Internet.

DETAILED DESCRIPTION:
Rates of obesity in the United States have increased dramatically over the past four decades. Although research studies have demonstrated that weight loss is achievable through lifestyle modifications, the maintenance of weight reduction beyond six months remains a challenge.

This study will examine the feasibility of a telehealth program for weight maintenance. Telehealth is the delivery of health related services to promote healthy behaviors through the innovative use of technology, without the need for travel. The telehealth program will be accessible at home through Internet-enabled television sets. The telehealth program includes three components: (1) weekly video programs that discuss problem solving and relapse prevention strategies and include motivational stories; (2) regularly updated video exercise programs; and (3) online communication with other study participants and an exercise and nutrition specialist.

A randomized controlled trial will determine the feasibility and acceptability of the weight maintenance telehealth program. The study participants will be African-American women, as they have a higher prevalence of obesity with a disproportionate risk of related chronic diseases (e.g., diabetes). Two churches will collaborate with the University of Illinois at Chicago and assist in meeting the social, spiritual, and cultural needs of the participants. One hundred women will be recruited to participate in a one-year trial. The study includes a weight loss phase (Phase 1), and a weight maintenance phase (Phase 2). During Phase 1, all participants will attend a 12-week weight loss program held in the participating churches. Following completion of this program, one church will be assigned to be the intervention group, and the other church will be the comparison group. During Phase 2, participants in the intervention group will receive monthly telephone counseling plus access to the telehealth program, while the comparison group will only receive monthly telephone counseling. The specific aims of the study include: (1) to evaluate the effect of the telehealth program on change in body mass index; and (2) to evaluate the effect of the telehealth program on physical activity and fat, fiber, fruit and vegetable intake.

ELIGIBILITY:
Inclusion Criteria:

* Self-identification as an African-American or Black woman
* Age 35-65 years
* Body mass index 25-50 kg/m2
* Physician approval to safely exercise if any positive answers on Physical Activity Readiness Questionnaire
* Owns a television
* Has a working telephone line

Exclusion Criteria:

* Plans to move from the Chicago area during the coming year
* Has a household member already in the study
* Uses illicit drugs or drinks more than two alcoholic drinks daily
* Pregnant, nursing, or planning pregnancy
* Participating in an organized weight loss program or using pharmacotherapy for weight loss
* Use an assistive device for ambulation, or cannot participate in exercise classes

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2007-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Body mass index | 12 months

SECONDARY OUTCOMES:
Physical activity | 12 months
Dietary intake | 12 months
  Dietary intake includes fat, fiber, fruits and vegetables.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Gerber, MD, MPH, Principal Investigator — University of Illinois at Chicago

REFERENCES:
- [Result] Gerber BS, Schiffer L, Brown AA, Berbaum ML, Rimmer JH, Braunschweig CL, Fitzgibbon ML. Video telehealth for weight maintenance of African-American women. J Telemed Telecare. 2013 Jul;19(5):266-72. doi: 10.1177/1357633X13490901. Epub 2013 Jun 14. PMID 24163236